CLINICAL TRIAL: NCT02505503
Title: Randomised Crossover Study With Nested Qualitative Component Investigating the Clinical Efficacy and Acceptability of Unloading Shoes in Patients With Intermittent Claudication Due to Peripheral Arterial Disease
Brief Title: York Study of Unloading Shoes for Vascular Intermittent Claudication
Acronym: YORVIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of York (Other); York St John University (Other); University of Salford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: YOR - A02382
Record Dates: First submitted 2015-07-15; First posted 2015-07-22 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Intermittent Claudication; Peripheral Arterial Disease
Keywords: Claudication; Footwear; Shoes; Walking capacity; Walking distance
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unloading shoes (Active Comparator): The unloading shoe will be a trainer-type shoe with a cosmetically-shaped rocker sole. The sole will have three circular curves whose arc centres are positioned at the anatomical ankle, hip and knee respectively; assuming a vertical lower limb. This is designed to influence the line of action of the ground reaction force to pass close to the anatomical joint centres and so reduce the moments needed to be generated for ambulation by the muscles acting across those joints in the lower limb. Additionally it is designed to place the ankle into a relatively plantarflexed position where the ankle plantarflexors use less energy than for instance when placed in dorsiflexion.
  Interventions: Device: Unloading shoes; Device: Unadapted control shoe
- Unadapted control shoes (Placebo Comparator): The control shoes will be similar in appearance to the unloading shoes, but they will not contain the altered sole.
  Interventions: Device: Unloading shoes; Device: Unadapted control shoe

INTERVENTIONS:
Device: Unloading shoes — The unloading shoe will be a trainer-type shoe with a rocker sole incorporated. The sole is designed to influence the line of action of the ground reaction force to pass close to the anatomical joint centres and so reduce the moments needed to be generated for ambulation by the muscles acting across those joints in the lower limb. Additionally it is designed to place the ankle into a relatively plantarflexed position where the ankle plantarflexors use less energy than for instance when placed in dorsiflexion.
Device: Unadapted control shoe — During the control condition assessments, participants wear a pair of appropriately-sized shoes, which are similar in appearance to the unloading shoes, but do not contain the altered sole.

SUMMARY:
Some people experience a cramp-like leg pain during walking that is relieved only by rest. This is called intermittent claudication (IC) and it is a common symptom of peripheral arterial disease. Patients with IC struggle to walk, which in turn lowers their quality of life.

The intensity of IC pain experienced during walking depends on several factors, including the type of footwear worn. For example, non-supportive shoes may make the calf muscles work harder during walking, leading to earlier and more-severe symptoms of IC.

A member of the research team has developed a shoe that reduces the work done by the lower-leg muscles during walking. Preliminary data indicate that, when wearing these "unloading shoes", people with IC were able to walk further without pain as compared with when wearing a normal pair of shoes. The current project aims to provide further information on the usefulness and acceptability of these shoes.

Forty people with IC will complete a set of three walking tests on two separate occasions; once whilst wearing the unloading shoes, and once whilst wearing some normal shoes. The participants will then be given a pair of unloading or normal shoes to wear for two weeks, after which we will collect information on how acceptable the shoes were to wear via a survey of all participants and one-to-one interviews with a subset of participants.

DETAILED DESCRIPTION:
Study design This is a single-centre, randomised crossover study with a qualitative component. Forty patients will be recruited from York Hospital. Participants will be asked to perform walking assessments on two week days within a maximum period of two weeks. Participants will be randomly assigned to complete walking assessments whilst wearing unloading shoes on day 1, followed by walking assessments whilst wearing control shoes on day 2, or vice versa. All participants will then be given the unloading or control shoes to wear for two weeks, after which they will complete a survey about how acceptable the shoes were to wear. A sub-sample of participants will also be interviewed about the acceptability of the shoes.

Study setting Recruitment for this study will take place at York Hospital, York, United Kingdom. Study assessments will take place at York St John University.

Unloading shoe The design of the "unloading" shoe to be used in this research will be a modern style of trainer-type shoe with a cosmetically-shaped rocker sole incorporated. The rocker sole will comprise of three circular curves whose arc centres are positioned at the anatomical ankle, hip and knee respectively; assuming a vertical lower limb. This is designed to influence the line of action of the ground reaction force to pass close to the anatomical joint centres and so reduce the moments needed to be generated for ambulation by the muscles acting across those joints in the lower limb. Additionally it is designed to place the ankle into a relatively plantarflexed position where the ankle plantarflexors use less energy than for instance when placed in dorsiflexion. This is in order to unload the calf muscles by providing a simultaneous reduction in ankle range of motion in relative plantarflexion but still moving with a near-normal trajectory. This also optimises the lever arm between the Achilles tendon and the ankle joint so making propulsion, and therefore calf muscle power generation, more efficient. Participants will be provided with a pair of appropriately-sized shoes, which will be produced for this study by an established shoe manufacturer - Chaneco (www.chaneco.co.uk). To allow participants to habituate to wearing the shoes before assessment, they will be allowed to walk around in the shoes at a self-selected pace for at least 5 minutes.

Control shoe During the control condition assessments, participants will wear a pair of appropriately-sized shoes, which are similar in appearance to the unloading shoes, but do not contain the altered sole. Again, these will be provided by Chaneco, and a minimum of 5 minutes walking will be allowed for habituation.

Outcome measures Primary outcome measure

• Maximum walking distance during forced-pace walking: Following a rest period of at least 20 minutes, participants will complete a 6-minute walk test in which they will be instructed to walk as far as possible within 6 minutes. This test simulates community walking better than treadmill testing, has been recommended as a primary outcome in claudication trials, and has good inter-day reproducibility (coefficient of variation 10.4%). A straight 30-m course will be used and the distance walked recorded. A testing checklist and standardised instructions will be used. The outcome assessor will have no role in the sizing and fitting of the shoes, in an attempt to keep them blinded, and the verbal test instructions will be audio-recorded so that we can check the consistency of which the instructions have been delivered.

Secondary outcome measures

* Pain-free walking distance during usual-pace walking: Following a rest period of at least 20 minutes, participants will be invited to walk at their usual walking speed along a straight 30-m course. Their walking speed will be recorded using electronic timing gates (SMARTSPEED, Fusion Sport). Participants will be instructed to indicate the point where they first experience claudication pain. The distance walked up until this point will be recorded.
* Gait biomechanical parameters: Reflective markers will be positioned on anatomical landmarks of the lower extremities using double-sided sticky tape to allow 3D motion analysis. Wireless surface electromyography units (Trigno EMG, Delsys, Italy) will also be attached to the skin overlying the medial and lateral Gastrocnemius and Tibialis Anterior using double-sided sticky tape to allow the assessment of lower-leg muscle recruitment patterns during the gait cycle. Participants will walk at their usual pace along a figure-of-8 circuit. A force plate (9281EA, Kistler) positioned in the central straight portion of the figure-of-8 will capture kinetic data. The participants will be naïve to the force plate, to help ensure a natural walking gait. Infra-red 3D optical motion analysis cameras (Oqus, Qualisys) will capture kinematic data each time a participant approaches and passes over the force plate. Participants will indicate when they experience the onset of claudication pain and continue until pain prevents them walking further. Outcomes include step length, stride length, cadence, velocity and joint angles, and joint moments and powers of the lower extremities during the three stages of pain development during walking; pain-free walking, after the onset of pain and immediately before stopping walking due to pain.

Participant timeline Participants will be required to attend the biomechanics laboratory at York St John University on 3 occasions: a first "screening" visit for obtaining written informed consent, confirming eligibility and recording baseline characteristics of the participant, and two subsequent visits on which the study assessments will be conducted. The study assessment sessions (i.e. visits 2 and 3) will be identical in composition apart from that the participants will wear different shoes (unloading or control) during the walking tests. The first assessment visit must be completed within 4 weeks of the screening visit, and there will be a maximum of 2 weeks and a minimum of 1 day between assessment visits 1 and 2. After completing the crossover study, half of the participants (n=20) will be given the unloading shoes and the other half (n=20) the control shoes to wear for 2 weeks. After this 2-week period, all participants will complete and return a survey about the shoes and be questioned via telephone about any adverse device effects. A sub-sample (minimum n=12; control n=6, unloading n=6) will undertake a telephone-based semi-structured interview with a qualitative researcher. This interview will be conducted within 2 weeks of the end of the 2 week shoe-wearing period. Therefore, the maximum duration that a participant will be involved in the study from the point of consenting is 10 weeks, and the minimum is 17 days; however, most participants will most likely be undertaking the study visits across a period of 4-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥16 years with intermittent claudication due to peripheral arterial disease
* Resting ankle-brachial index ≤0.9 and/or imaging evidence of peripheral arterial disease
* Stable symptoms for at least 3 months (assessed via self-report)
* Pain-free walking distance <250 m on 6-minute walk test
* Ambulation that is limited primarily by calf claudication on 6-minute walk test
* Able to provide written informed consent
* Able to read and speak English

Exclusion Criteria:

* Absolute contraindications to exercise testing as defined by the American College of Sports Medicine
* Critical limb ischemia
* Function is uniquely impaired, e.g. vascular amputees
* Co-morbidities that limit walking to a greater extent than intermittent claudication (e.g. severe arthritis)
* Ambulation limited by claudication in regions other than the calf
* Current or previous (within 6 months) use of shoe inserts, knee or ankle braces or customised shoes prescribed by a health professional
* Ankle/foot pathology/pain on either side
* "High-risk" foot (e.g. significant peripheral neuropathy, foot deformity, history of foot ulceration), assessed by a vascular specialist (Registrar or Consultant) or podiatrist

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Total distance walked during 6-minute walk test | Measured 40 minutes after putting on the intervention or control shoes
  Following a rest period of at least 20 minutes, participants will complete a 6-minute walk test in which they will be instructed to walk as far as possible within 6 minutes. A straight 30-m course will be used and the distance walked recorded.

SECONDARY OUTCOMES:
Pain-free walking distance during usual-pace walking | Measured 20 minutes after putting on the intervention or control shoes
  Following a rest period of at least 20 minutes, participants will be invited to walk at their usual walking speed along a straight 30-m course. Participants will be instructed to indicate the point where they first experience claudication pain. The distance walked up until this point will be recorded.
Walking speed | Measured 60 minutes after putting on the intervention or control shoes
  This variable will be assessed during self-paced walking.
Step length | Measured 60 minutes after putting on the intervention or control shoes
  This variable will be assessed during self-paced walking.
Step cadence | Measured 60 minutes after putting on the intervention or control shoes
  This variable will be assessed during self-paced walking.
Muscle activation | Measured 60 minutes after putting on the intervention or control shoes
  Electromyography will be used to observe when during the gait cycle of self-paced walking the calf muscles are activated. This will allow the investigators to determine the effectiveness of the unloading shoes in altering calf muscle activity.
Joint moments | Measured 60 minutes after putting on the intervention or control shoes
  An infrared camera system and force platform will be used to assess external moments at the ankle, knee and hip.

OTHER OUTCOMES:
Adverse events / adverse device effects | Participants will be followed for the duration of their study involvement, an expected average of 5 weeks.
  For the purpose of this study the adverse events that will be recorded are those that may occur as a result of performing any of the study assessments (e.g. walking tests), or the use of the study shoes (i.e. the investigational device).

CONTACTS AND LOCATIONS:
Overall Officials: Garry Tew, PhD, Principal Investigator — University of York
Locations (2):
- United Kingdom (2):
  - York St John University, York, North Yorkshire
  - York Teaching Hospital NHS Foundation Trust, York, North Yorkshire

REFERENCES:
- [Derived] Jordan AR, Tew GA, Hutchins SW, Shalan A, Cook L, Thompson A. Three-curve rocker-soled shoes and gait adaptations to intermittent claudication pain: A randomised crossover trial. Gait Posture. 2019 Jan;67:31-36. doi: 10.1016/j.gaitpost.2018.09.001. Epub 2018 Sep 22. PMID 30265963
- [Derived] Tew GA, Shalan A, Jordan AR, Cook L, Coleman ES, Fairhurst C, Hewitt C, Hutchins SW, Thompson A. Unloading shoes for intermittent claudication: a randomised crossover trial. BMC Cardiovasc Disord. 2017 Nov 28;17(1):283. doi: 10.1186/s12872-017-0716-x. PMID 29179693